CLINICAL TRIAL: NCT06977152
Title: Comparison of the Effectiveness of Fluidized Positioner and Memory Foam Pillow in the Prevention of Pressure Injury in the Children's Head: A Randomised Controlled Study
Brief Title: Comparison of the Effectiveness of Fluidized Positioner and Memory Foam Pillow in the Prevention of Pressure Injury in the Children's Head
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Koç University (Other)
Collaborators: Koç University Hospital (Unknown)
Responsible Party: Principal Investigator, Enes Simsek, Principal Investigator, Koç University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2025.114.IRB2.059
Record Dates: First submitted 2025-04-26; First posted 2025-05-18 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-05

CONDITIONS: Pressure Injury
Keywords: pediatric patients; Pressure injury; Risk assessment; foam pillow; fluidized positioner
MeSH Terms: conditions — Pressure Ulcer

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fluidized positioner (Experimental): Patients in the experimental group will have a fluidized positioner placed under their head and neck immediately after the initiation of mechanical ventilation support in the PICU.
  Interventions: Device: Fluidized Positioner
- Memory foam pillow (Active Comparator): Patients in the comparison group will have a memory foam pillow placed under their head and neck immediately after the initiation of mechanical ventilation support in the PICU.
  Interventions: Device: Memory foam pillow

INTERVENTIONS:
Device: Memory foam pillow — Patients in the memory foam pillow intervention group will have a memory foam pillow placed under their head and neck immediately after the initiation of mechanical ventilation support in the PICU.
  Arms: Memory foam pillow
Device: Fluidized Positioner — Patients in the fluidized positioner intervention group will have a fluidized positioner placed under their head and neck immediately after the initiation of mechanical ventilation support in the PICU.
  Arms: Fluidized positioner

SUMMARY:
This study aims to compare the effectiveness of fluidized positioners and memory foam pillows in preventing pressure injuries in the head among pediatric patients.

H1: There is a significant difference between the fluidized positioner and the memory foam pillow in terms of pressure injury incidence in pediatric intensive care patients.

H2: The fluidized positioner reduces the risk of developing pressure injuries more effectively than the memory foam pillow.

H3: There is a significant difference in the pressure applied to the head region of the patient between the fluidized positioner and the memory foam pillow.

H4: The anatomical locations of pressure injuries (occipital, parietal, temporal, and ear regions) vary depending on the type of pillow used.

H5: Compared to the memory foam pillow, the fluidized positioner provides a more evenly distributed pressure across the occipital, parietal, temporal, and ear regions and prevents pressure concentration in specific areas.

ELIGIBILITY:
Inclusion Criteria:

* Being treated in the pediatric intensive care unit
* Being mechanically ventilated
* Being immobile, being in age interval of 28 days to 5 years
* Having consent for the participation of the study

Exclusion Criteria:

* Having surgical intervention in the head region
* Parents want to leave at any stage of the project
* Having hydrocephalus or burn in the head area
* Having PIs on admission to hospital
* Existing dermatologic diseases affecting the skin or connective tissue
* Having emergence of a new condition during the intervention may significantly affect the risk of pressure injury (e.g., sudden surgery or complication)
* Inability to obtain sufficient data during the study (e.g., patient transfer)

Ages: 28 Days to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 64 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Pressure Injury Development | 0-14 days after the beginning of mechanical ventilation support
  The study will compare the incidence, stage, and anatomical location of PIs between the two groups.

SECONDARY OUTCOMES:
Pressure Measurement | At multiple time points in the 0-14th day after beginning of mechanical ventilation support
  Interface pressure will be evaluated using a circular-shaped pressure sensor specialized for this measurement.

CONTACTS AND LOCATIONS:
Overall Officials: Enes Şimşek, MSc. PhD(c), Principal Investigator — Koç University
Locations (1):
- Koç University Hospital, Istanbul, Zeytinburnu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No